CLINICAL TRIAL: NCT04415840
Title: Benefits of Using Lugol's Solution in Addition to Acetic Acid During Colposcopy in Women With Cervical Dysplasia
Brief Title: Lugol's Solution in Addition to Acetic Acid During Colposcopy
Status: Completed | Type: Observational
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Sponsor
Other Study IDs: COLPO-4
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-04

CONDITIONS: Uterine Cervical Dysplasia
Keywords: cervical dysplasia; colposcopy; Lugol's solution; acetic acid
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: acetic acid test — using acetic acid to unmask dysplastic lesions on the cervix uteri
Diagnostic Test: Lugol's solution test — using Lugol's solution after acetic acid test to unmask dysplastic lesions on the cervix uteri

SUMMARY:
To assess the benefits of using Lugol's solution in addition to acetic acid during colposcopy in women with cervical dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* women referred for colposcopy due to cervical abnormalities
* written informed consent

Exclusion Criteria:

* pregnant women
* presence of a language barrier
* history of conization or other treatments on the cervix uteri
* iodine allergy

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Non-pregnant women referred for colposcopy due to cervical abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
additional identified dysplastic lesions on the cervix uteri due to the use of Lugol's Solution | 1 minute
  We count all the cases in which dysplastic lesions on the cervix uteri where identified due to the use

SECONDARY OUTCOMES:
Sensitivity | 1 minute
  sensitivity of the examination (acetic acid + Lugol´s solution)
Specificity | 1 minute
  Specificity of the examination (acetic acid + Lugol´s solution)
PPV | 1 minute
  Positive predictive value of the examination (acetic acid + Lugol´s solution)
NPV | 1 minute
  Negative predictive value of the examination (acetic acid + Lugol´s solution)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (2):
- Germany (2):
  - Zydolab - Institute of Cytology and Immune Cytochemistry, Dortmund, North Rhine-Westphalia
  - Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No